CLINICAL TRIAL: NCT02868801
Title: Efficacy and Safety of Pregabalin Sustained Release Tablet for Postherpetic Neuralgia -A Multicenter,Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Pregabalin Sustained Release Tablet for Postherpetic Neuralgia
Acronym: EASOPSRTFP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRPRBL-PHN
Record Dates: First submitted 2015-07-08; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-02

CONDITIONS: Postherpetic Neuralgia
Keywords: Pregabalin
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): placebo, oral administration for 14 weeks (2 week titration and 12-week fixed dose)
  Interventions: Drug: Placebo
- Pregabalin SR tablet 165mg/day (Experimental): 1pills once ,one time a day in an hour after meals, oral administration for 14 weeks (2 week titration and 12-week fixed dose)
  Interventions: Drug: Pregabalin SR tablet 165mg/day
- Pregabalin SR tablet 330mg/day (Experimental): 1pills once ,one time a day in an hour after meals, oral administration for 14 weeks (2 week titration and 12-week fixed dose)
  Interventions: Drug: Pregabalin SR tablet 330mg/day
- Pregabalin SR tablet 660mg/day (Experimental): 2pills once ,one time a day in an hour after meals, oral administration for 14 weeks (2 week titration and 12-week fixed dose)
  Interventions: Drug: Pregabalin SR tablet 660mg/day

INTERVENTIONS:
Drug: Placebo — same intervention as the experimental group
  Other Names: Placebo tablet of pregabalin sustained release tablet
  Arms: Placebo
Drug: Pregabalin SR tablet 165mg/day — According to the efficacy and safety in titration
  Other Names: Pregabalin sustained release tablet
  Arms: Pregabalin SR tablet 165mg/day
Drug: Pregabalin SR tablet 330mg/day — According to the efficacy and safety in titration
  Other Names: Pregabalin sustained release tablet
  Arms: Pregabalin SR tablet 330mg/day
Drug: Pregabalin SR tablet 660mg/day — According to the efficacy and safety in titration.
  Other Names: Pregabalin sustained release tablet
  Arms: Pregabalin SR tablet 660mg/day

SUMMARY:
The purpose of this study is to evaluate the Efficacy and safety of pregabalin sustained release tablet versus placebo for postherpetic neuralgia.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicenter, placebo-controlled trial to compare the efficacy and safety of pregabalin SR vs placebo in patients with PHN.

The study is conducting at 27 study centers in China. Patients were randomized to receive pregabalin, starting at 165 mg/day and increasing to a maintenance dose of 330 or 660 mg/day, or placebo.

The study includes a 1-week, single-blind, placebo run-in period; a 2-week dose-escalation/optimization phase; a 12-week, fixed-dose treatment period; and a 1-week taper phase.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient ，Patients can not stay in the hospital overnight；
2. Patients must have pain present for more than 3 months after the healing of the herpes zoster skin rash；
3. At least 4 days and at least 8 pain diaries(Pain Numeric Rating Scale) must be completed satisfactorily within the seven days of single-blind, placebo run-in period, and the average pain score must be greater than or equal to 4；
4. At screening (V0) and enrollment (V1), patients must have a score of greater than or equal to 40 mm on the 100 mm pain visual analog scale；
5. Women were neither pregnant nor lactating, and those of childbearing age had a confirmed negative serum pregnancy test at baseline and practiced an appropriate method of contraception throughout the study.

Exclusion Criteria:

1. Decrease of ≥30% on their pain VAS or ≥ 4 between any two pain diaries during the placebo run-in period.( in order to remove potential placebo-responders)；
2. Patients who had failed to respond to previous treatment for PHN with gabapentin at doses ≥1200 mg/day ；
3. History of using pregabalin or participation in a previous trial of pregabalin；
4. Patients with a skin condition or severe non-PHN pain that might impair the self assessment of pain caused by PHN；
5. Patients with other Nervous system disorders which might impair completing the pain diaries or sleep interference diaries；
6. History of epilepsy and being treated by drug therapy；
7. Previous surgical therapy for PHN；
8. History of using effective therapies during 2 weeks before screening (V0),eg: acupuncture and moxibustion, Transcutaneous Electrical Nerve Stimulation；
9. Potentially retinal toxicity of drugs past or now；
10. Prohibited medications without appropriate washout；
11. Malignancy within the past 2 years；
12. Laboratory examination: WBC<2.5×109/L；ANC<1.5×109/L；PLT<100×109/L；ALT/AST>3ULN；
13. Creatinine clearance ≤ 60 mL/min；
14. Positive antibody of Hepatitis c，Human immunodeficiency virus ，Treponema pallidum ；
15. Patients who are allergic to or intolerant of pregabalin or other drugs which have a similarly chemical structure ；
16. History of illicit drug or alcohol abuse within the last 2 years；
17. Clinically significant or unstable hepatic, respiratory, or hematologic illnesses or psychologic conditions; unstable cardiovascular disease which may increase the risk of participation the clinical trial in the opinion of the study investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of Responders | 15 weeks
  A responder is defined as a subject with a 30% reduction in weekly mean pain score from baseline to endpoint

SECONDARY OUTCOMES:
50% reduction in weekly mean pain score from baseline to study completion | 15 weeks
Change of Mean Pain Scores from study completion to baseline | 15 weeks
Change of Mean Sleep Interference Scores from study completion to baseline | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lu Qianjin, M.D., Principal Investigator — Second Xiangya Hospital of Central South University
Locations (27):
- China (27):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chao-yang Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-Sen Memory Hospital , Sun Yat-Sen University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - Fourth Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital Of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Yancheng City NO.1 People's Hospital, Yancheng, Jiangsu
  - The Affiliated Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital Of China Medical University, Shengyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Qingdao Municipal Hospital(Group), Qingdao, Shandong
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital Of Shanxi Medical University, Taiyuan, Shanxi
  - Second Hospital Of Shanxi Medical University, Taiyuan, Shanxi
  - Xijing Hospital; the Fourth Military Medical University, Xi’an, Shanxi
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Xinjiang Uygur Autonomous Region Hospital OF TCM, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital , Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] van Seventer R, Feister HA, Young JP Jr, Stoker M, Versavel M, Rigaudy L. Efficacy and tolerability of twice-daily pregabalin for treating pain and related sleep interference in postherpetic neuralgia: a 13-week, randomized trial. Curr Med Res Opin. 2006 Feb;22(2):375-84. doi: 10.1185/030079906x80404. PMID 16466610